CLINICAL TRIAL: NCT03305718
Title: Biomarkers of Meats and Potatoes Intake: a Meal Study in Healthy Men and Women - the MEPO Study.
Brief Title: Biomarkers of Meats and Potatoes Intake.
Acronym: MEPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-15020401
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Biomarkers of Food Intake in Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Meal sequence: 3C1A2B4D (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 3C1A2B4D.
  Interventions: Other: Meal sequence: 3C1A2B4D
- Meal sequence: 2A3D4C1B (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 2A3D4C1B.
  Interventions: Other: Meal sequence: 2A3D4C1B
- Meal sequence: 2D4B3A1C (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 2D4B3A1C.
  Interventions: Other: Meal sequence: 2D4B3A1C
- Meal sequence: 3B2C1D4A (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 3B2C1D4A.
  Interventions: Other: Meal sequence: 3B2C1D4A
- Meal sequence: 4C2B1A3D (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 4C2B1A3D.
  Interventions: Other: Meal sequence: 4C2B1A3D
- Meal sequence:1B4D3C2A (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 1B4D3C2A.
  Interventions: Other: Meal sequence:1B4D3C2A
- Meal sequence:4A1C2D3B (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 4A1C2D3B.
  Interventions: Other: Meal sequence:4A1C2D3B
- Meal sequence:1D3A4B2C (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 1D3A4B2C.
  Interventions: Other: Meal sequence:1D3A4B2C
- Meal sequence: 4D3B2C1A (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 4D3B2C1A.
  Interventions: Other: Meal sequence: 4D3B2C1A
- Meal sequence: 3A4C1B2D (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 3A4C1B2D.
  Interventions: Other: Meal sequence: 3A4C1B2D
- Meal sequence: 1C2A3D4B (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 1C2A3D4B.
  Interventions: Other: Meal sequence: 1C2A3D4B
- Meal sequence: 2B1D4A3C (Experimental): In this study, each participant was randomized to a sequence of the 4 meat meals and to a sequence of the 4 potato meals. The four meat meals consist of a beef meal, a pork meal, a chicken meal or a control meal (1-4). The four potato meals consist of french fries, chips, boiled potatoes or rice (A-D). The test meal consists of one meat meal that was served together with a potato meal. Four different test meals were served in four interventions, separated by a washout period of minimum 12 days. Six hours after the test meal an ad libitum meal was served, consisting of vegetable stew with pasta.
  Each participants randomized to this arm is exposed to 4 test meals in the order 2B1D4A3C.
  Interventions: Other: Meal sequence: 2B1D4A3C

INTERVENTIONS:
Other: Meal sequence: 3C1A2B4D — Participants receive test meals in the sequence 3C1A2B4D
  Arms: Meal sequence: 3C1A2B4D
Other: Meal sequence: 2A3D4C1B — Participants receive test meals in the sequence 2A3D4C1B
  Arms: Meal sequence: 2A3D4C1B
Other: Meal sequence: 2D4B3A1C — Participants receive test meals in the sequence 2D4B3A1C
  Arms: Meal sequence: 2D4B3A1C
Other: Meal sequence: 3B2C1D4A — Participants receive test meals in the sequence 3B2C1D4A
  Arms: Meal sequence: 3B2C1D4A
Other: Meal sequence: 4C2B1A3D — Participants receive test meals in the sequence 4C2B1A3D
  Arms: Meal sequence: 4C2B1A3D
Other: Meal sequence:1B4D3C2A — Participants receive test meals in the sequence 1B4D3C2A
  Arms: Meal sequence:1B4D3C2A
Other: Meal sequence:4A1C2D3B — Participants receive test meals in the sequence 4A1C2D3B
  Arms: Meal sequence:4A1C2D3B
Other: Meal sequence:1D3A4B2C — Participants receive test meals in the sequence 1D3A4B2C
  Arms: Meal sequence:1D3A4B2C
Other: Meal sequence: 4D3B2C1A — Participants receive test meals in the sequence 4D3B2C1A
  Arms: Meal sequence: 4D3B2C1A
Other: Meal sequence: 3A4C1B2D — Participants receive test meals in the sequence 3A4C1B2D
  Arms: Meal sequence: 3A4C1B2D
Other: Meal sequence: 1C2A3D4B — Participants receive test meals in the sequence 1C2A3D4B
  Arms: Meal sequence: 1C2A3D4B
Other: Meal sequence: 2B1D4A3C — Participants receive test meals in the sequence 2B1D4A3C
  Arms: Meal sequence: 2B1D4A3C

SUMMARY:
The discovery of biomarkers for the intake of meats and potatoes is needed for an accurate assessment of the intake of these foods. Twelve healthy subjects were enrolled in a controlled, cross-over meal study, randomized by a Latin square design. The test meals contained 1) beef, pork, chicken and a control meal for the meats and 2) french fries, boiled potatoes, chips and a control for the potato meals. A standardized diet was provided during sample collection. Blood and urine samples were collected up to 48h primarily for untargeted metabolomic profiling. Blood was further collected to study the effect of the meals on insulin and glycemic responses. Effects on satiety were measured by VAS and an ad libitum lunch following the test meals.

DETAILED DESCRIPTION:
Protein-rich diets improve body weight regulations and are thus believed to play a key role in combating the global obesity epidemic. Protein-rich diets are generally high in meats, some of which have become controverted enough to be considered disease-promoting foods despite their nutritional richness. The degree at which associations with disease differs from causality is however not entirely known.

Assessment of food intake currently relies on food frequency questionnaires (FFQ), 24h recall and dietary records, all of which are self-reporting methods known to be subject to bias and inaccuracy. Biomarkers of food intake emerged thus within the past years to complement the conventional tools as objective measurements of food intake, drawn from biological samples. Several biomarkers of meat consumption have been proposed, however none is currently accepted and used as biomarker(s) of meat intake and none is able to differentiate between the different types of meat.

In the modern diet, meats are very often served with potatoes. To our knowledge, biomarkers of potato intake have not been thoroughly reported in the literature. Different cooking methods were shown to potentially influence the content of bioactive constituents of vegetables, their glycemic index, as well as subsequent energy intake. High heat cooking additionally yields the formation of potentially toxic compounds such as advanced glycation endproducts (AGEs) that were shown to contribute to insulin resistance and type 2 diabetes. In this line, biomarkers of potatoes as such as well as biomarkers to differentiate between different cooking methods would be of great importance in advancing the understanding of nutritional science.

Primary objectives:

1. To identify acute biomarkers of general meat intake by untargeted metabolomics
2. To explore the changes in the metabolome as a result of acute exposure to three types of meat and identify meat-specific biomarkers of intake
3. To identify biomarkers of acute potato intake by untargeted metabolomics
4. To identify biomarkers that can differentiate between three types of cooking methods
5. To investigate the effect of the interaction between meat on potatoes on satiety, assessed by registration of intake from an ad libitum meal

Secondary objectives:

1. To validate already known biomarkers of meat intake by targeted metabolomics
2. To investigate the effect of the interaction between meat and potatoes on satiety, assessed by visual analogue scales
3. To investigate the effect of the interaction between meat and potatoes on glucose and insulin responses

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30 kg/m2
* Eating and tolerating meat, egg, pea, rice, and potatoes
* No current chronic or infectious disease
* No medication (oral contraceptive pill and mild antidepressants is allowed)
* No dietary supplements
* Did not use antibiotics in the 6 previous months

Exclusion Criteria:

* Any condition that makes the project responsible researcher to doubt the feasibility of the volunteer's participation
* Pregnant or lactating women
* Smoking (12 months of non-smoking is allowed)
* Vegan or vegetarian
* Have or have had a drug addiction
* Blood donations within three months before participating in the current trial or participation in other scientific experiments
* Alcohol consumption higher than the Danish Health Authority recommendation of 7 or 14 drinks/week for women and men, respectively.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Urinary meat metabolites (metabolic profiling with mass spectrometry) | Hours 0-48
  Explorative approach to discover biomarkers of general meat intake and to differentiate between different types of meat
Plasma meat metabolites (metabolic profiling with mass spectrometry) | Hours 0-48
  Explorative approach to discover biomarkers related to general meat intake and/or specific types of meat
Urinary potato metabolites (metabolic profiling with mass spectrometry) | Hours 0-48
  Explorative approach to discover biomarkers of general potato intake and to differentiate between different cooking methods
Plasma potato metabolites (metabolic profiling with mass spectrometry) | Hours 0-48
  Explorative approach to discover biomarkers related to general potato intake and/or related to different cooking methods
Objective assessment of satiety | Hours 0-7
  Measured by the weight of an ad libitum meal

SECONDARY OUTCOMES:
Urine biomarkers of meat intake | Hours 0-48
  Targeted approach with mass spectrometry on already proposed meat biomarkers
Subjective assessment of satiety | Hours 0-6
  Assessed by visual analogue scale (VAS)
Area under the curve for glucose | Minutes 0-180
  Glucose is measure at 0, 45, 90, 120, and 180 min after the test meal and the area is determined by the trapezoid method.
Area under the curve for insulin | Minutes 0-180
  Insulin is measure at 0, 45, 90, 120, and 180 min after the test meal and the area is determined by the trapezoid method.